CLINICAL TRIAL: NCT02883907
Title: Advanced MR Imaging of Osteoarthritis
Acronym: AMROA
Status: Completed | Type: Observational
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Jamie MacKay, Clinical Research Fellow, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: 609/M/C/1670
Record Dates: First submitted 2016-08-22; First posted 2016-08-30 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples for cartilage turnover marker measurement

GROUPS / COHORTS (2):
- Healthy volunteers
- Osteoarthritis patients

SUMMARY:
The utility of conventional imaging in the development of new treatments for osteoarthritis (OA) is hindered by:

1. Difficulty in non-invasively evaluating the initial response to potential new treatment options. OA typically develops over a long time period, so evaluating the efficacy of new treatment options over a timeframe relevant to experimental medicine studies is difficult.
2. Inadequate methods of disease quantification and stratification. OA is a heterogeneous condition and identifying which subgroups of patients are most likely to benefit from new treatments is crucial.

Novel magnetic resonance (MR) imaging acquisition and analysis techniques have the potential to solve these problems. However, their reliability needs to be fully established and knowledge of likely effect sizes is required to inform sample size considerations for further longitudinal/interventional studies.

This study aims to help address these issues by:

1. Calculating effect sizes for MR measurements to inform sample size calculations for future studies.
2. Assessing the reliability of a multiparametric MR protocol for assessment of the knee joint.

The investigators will examine a single knee of an initial 15 participants with MR. Participants will be drawn from two groups: (1) 10 participants aged 40-60 years old with clinical and x-ray features of OA and (2) 5 control subjects (matched to cases for age, sex and body mass index in a 1:2 ratio) who do not have clinical features of OA.

Participants will undergo an initial (baseline) MR examination, followed by repeat MR examinations at approximately 1 month and 1 year following the baseline examination.

This will allow us to assess both the reliability of our MR measurements and the expected progression in our MR measurements in OA subjects in the absence of any disease-modifying intervention.

ELIGIBILITY:
Group 1 Inclusion Criteria:

* Meets American College of Rheumatology (ACR) criteria for OA
* Kellgren-Lawrence grade 2-3 OA on knee radiograph
* Medial compartment predominant disease
* Neutral alignment
* Aged 40-60
* Body Mass Index (BMI) < 35 kg per square meter
* Ambulatory and in good general health

Group 2 Inclusion Criteria:

* No current symptoms of knee pain or stiffness or other clinical features of OA
* Aged 40-60
* BMI < 35 kg per square meter
* Ambulatory and in good general health

Exclusion Criteria (both groups):

* History of ipsilateral lower limb fracture
* History of ipsilateral lower limb surgery (including arthroscopy)
* Metabolic bone disease
* Inflammatory arthritis
* Haematological malignancy
* Paget's disease
* Bone metastases
* Contraindication to MR imaging (e.g. pacemaker, severe claustrophobia)
* Contraindication to intravenous gadolinium based contrast medium administration (see 'Ethical Considerations' section)
* Unable to consent

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Group 1 will consist of 10 patients aged 40-60 who have presented to the Orthopaedic clinic with a painful knee, and have mild/moderate OA on plain radiographs (Kellgren-Lawrence grade 2-3).
  Group 2 will consist of 5 healthy volunteer controls, matched (1:2 ratio) to cases for age, sex and body mass index who do not have knee pain.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Mean cartilage T1rho relaxation time (milliseconds) | 1 year
Mean cartilage T2 relaxation time (milliseconds) | 1 year
Mean cartilage T1 relaxation time post gadolinium (milliseconds) | 1 year
  Derived from delayed gadolinium enhanced MR of cartilage (dGEMRIC)

SECONDARY OUTCOMES:
Modified Osteoarthritis Knee Score (MOAKS) (arbitrary units) | 1 year
  Semiquantitative scoring system
Cartilage thickness values (millimeters) | 1 year
  Surface-based comparison using statistical parametric mapping
Subchondral bone area (millimeters squared) | 1 year
Dynamic contrast enhanced (DCE) quantitation of parameters | 1 year
  Multiple DCE parameters calculated allowing description of enhancement rate and pattern of synovium
Subchondral bone texture index (arbitrary units) | 1 year
Osteochondral junction integrity (semiquantitative grading, arbitrary units) | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Addenbrooke's Hospital, Cambridge, Cambridgeshire, United Kingdom